CLINICAL TRIAL: NCT03309436
Title: Effects of Clomiphene Citrate Ovulation Induction on Frozen Embryo Transfer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIAI E2017-11
Record Dates: First submitted 2017-02-28; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-08

CONDITIONS: Infertility, Female; Clomiphene Citrate
MeSH Terms: conditions — Infertility, Female | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use Clomiphene Citrate protocol (Experimental): Ovulation induction: regular Clomiphene Citrate protocol. Start use rFSH or HMG from day 2/3 of the menstrual cycle, the initial dosage is determined by patients' age, BMI, antral follicle number, FSH, E2, AMH and past ovarian response, usually 150-225IU/d, until hCG injection. At the same time, take CC 100mg/d until hCG injection. The dosage of Gn will be adjust by serum E2, P, LH and the development of follicular.
  Interventions: Drug: Clomiphene Citrate protocol
- Procedure (Active Comparator): Ovulation induction: regular GnRH antagonist protocol. Start use rFSH or HMG from day 2/3 of the menstrual cycle, the initial dosage is determined by patients' age, BMI, antral follicle number, FSH, E2, AMH and past ovarian response, usually 150-225IU/d, until hCG injection. When a dominant follicle diameter over 14mm or serum E2 over 350pg/ml, use GnRH-ant 0.25mg/d, until hCG injection. The dosage of Gn will be adjust by serum E2, P, LH and the development of follicular.
  Interventions: Procedure: Procedure

INTERVENTIONS:
Drug: Clomiphene Citrate protocol — Take CC 100mg/d at the same time with Gn until hCG injection.
  Other Names: CC
  Arms: Use Clomiphene Citrate protocol
Procedure: Procedure — When a dominant follicle diameter over 14mm or serum E2 over 350pg/ml, use GnRH-ant 0.25mg/d, until hCG injection.
  Other Names: GnRH antagonist protocol
  Arms: Procedure

SUMMARY:
Clomiphene citrate has been widely used for treatment of infertility for decades. Although its anti-estrogenic effects leads to low pregnancy rate, clomiphene citrate is still a first-line treatment for ovulation induction because of its simple usage, low prices, no injection and low risk of ovarian hyperstimulation syndrome. Clomiphene citrate shows high affinity with estrogen receptor, which inhibits endometrial proliferation, inevitably leads to a decline in endometrial receptivity, thus affecting the success rate of IVF.

In that case, use clomiphene citrate for ovulation induction is lost more than gained based on fresh embryo transfer. But recently, some researchers have proposed to extend the time from ovulation induction to embryo transfer, and the increased level of estradiol can replace clomiphene citrate to combine with the receptor, so that the uterine environment is more conducive to pregnancy. Therefore, use clomiphene citrate based on vitrification of embryo maybe a good way for treatment of infertility.

At present, using frozen embryo transplantation after ovulation induction by clomiphene citrate is a common treatment, but few research has mentioned the best time for embryo implantation. The investigators research is to find the most appropriate time for frozen embryo implantation after using clomiphene citrate for ovulation induction.

DETAILED DESCRIPTION:
This study receives patients from 2017 August to 2018 June who undergo ART treatment at Shanghai Jiai Genetics & IVF Institute and taken either CC or GnRH antagonist protocol(control group) for ovulation induction.

The investigators will record every patients' age, BMI, serum E2, P, LH level, infertility factors and pregnancy outcomes, counted the implantation rate and clinical pregnancy rate, and then used SPSS Software x2 test for statistical analysis, the significance was set at p<0.05.The investigators will also make a correlation analysis about the serum hormone level and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

Women 18-40 years of age who are scheduled for IVF or ICSI in our IVF institute while meeting the following criteria:

1. AMH ≥ 2;
2. Infertility factors: tubal factor, severe oligospermia, etc;
3. FET cycle;
4. Cleavage stage embryo transfer (Day 3).

Exclusion Criteria:

1. BMI ≤ 18.4 or ≥ 25.0;
2. Have pregnancy complications;
3. Genital tract malformations, uterine cavity diseases, PCOS;
4. Endometriosis;
5. Genetic diseases, severe somatic diseases, mental disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | 4 weeks after embryo transfer for the patient
  Clinical pregnancy is defined as the presence of a gestational sac confirmed by transvaginal ultrasound examination.
  Clinical pregnancy rate per treatment cycle will also be calculated based on ITT.

SECONDARY OUTCOMES:
Ongoing pregnancy | 12 weeks after embryo transfer for the patient
  Ongoing pregnancy is defined as a viable intrauterine pregnancy after 12 weeks of embryo transfer. Ongoing pregnancy rate per treatment cycle will also be calculated on intend-to-treat(ITT) basis.
Implantation of transferred embryo | 2 weeks after embryo transfer for the patient
  Implantation rate per embryo transferred will also be calculated.

OTHER OUTCOMES:
Regression analysis 1 | 12 weeks after embryo transfer for the patient
  Regression analysis about the pregnancy outcomes and patients' serum E2,P4,LH levels on the day of hCG injection
Regression analysis 2 | 12 weeks after embryo transfer for the patient
  Regression analysis about the pregnancy outcomes and patients' serum E2,P4,LH levels on the day of embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, MD, Study Chair — Shanghai Jiai Genetics & IVF Institute
Locations (1):
- Shanghai Jiai Genetics & IVF Institute, Shanghai, China